CLINICAL TRIAL: NCT06619509
Title: A Phase II, Single-arm, Open-label, Long-term Safety Rollover Trial of Oral Brigimadlin in Patients With Solid Tumours
Brief Title: A Study to Test Long-term Treatment With Brigimadlin in People With Solid Tumours Who Took Part in a Previous Study With This Medicine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0032; 2024-514177-21-00 (Registry Identifier: CTIS); U1111-1305-3484 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumours
MeSH Terms: interventions — brigimadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brigimadlin (Experimental)
  Interventions: Drug: Brigimadlin

INTERVENTIONS:
Drug: Brigimadlin — Brigimadlin
  Other Names: BI 907828

SUMMARY:
This study is open to adults with solid tumours who received at least 4 cycles of treatment with brigimadlin in a previous study. The goal of this study is to find out how well people with solid tumours tolerate long-term treatment with brigimadlin. Brigimadlin is a so-called MDM2 inhibitor that was being developed to treat cancer.

All participants take brigimadlin as tablets once every 3 weeks at the study site. At study visits, doctors check participants' health and take note of any unwanted effects. At some study visits, doctors also check the size of the tumour and whether it has spread to other parts of the body. Participants are in the study as long as they benefit from treatment and can tolerate it.

ELIGIBILITY:
Inclusion criteria:

1. Patient is ongoing on brigimadlin treatment in any trial sponsored by Boehringer Ingelheim (hereafter referred to as the 'parent trial').
2. Provision of signed and dated, written informed consent form (ICF) in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
3. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use 2 medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of <1% per year when used consistently and correctly beginning at Screening, during trial participation, and until 6 months and 12 days after the last dose for women and 102 days after the last dose for men. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information.
4. Participants must be willing and able to comply with the scheduled visits, treatment plan, lifestyle, laboratory tests, contraceptive guidelines, and other study procedures.
5. Adequate organ function.
6. Patient is eligible to receive continued treatment according to the clinical trial protocol of the parent trial they are currently participating in. Patients currently experiencing a dose delay in the parent trial due to adverse events are eligible if recovery from the adverse event takes place within the allowed time window in the parent trial.

Exclusion criteria:

1. Any medical condition which in the opinion of the investigator should exclude the patient from receiving treatment with brigimadlin.
2. Participants who must receive or intend to receive restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
3. Women who are pregnant, nursing, or who plan to become pregnant while in the trial. Female patients who do not agree to the interruption of breastfeeding from the start of study treatment until 6 months and 12 days after the last dose of study treatment.
4. Patient has unacceptable toxicity on brigimadlin at the time of transition into this trial.
5. Patient has an adverse event (AE) which has caused a dose delay and has not recovered within the allowed time window in the parent trial.
6. Patient who has already required 2 dose reductions and would require a third dose reduction at trial entry, unless the investigator deems treatment continuation beneficial, and the third dose reduction is agreed in writing between the investigator and the sponsor.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the occurrence of treatment-emergent adverse events (AEs) according to CTCAE Version 5.0 during the entire treatment period | up to 9 years.
  CTCAE=Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Locations (50):
- United States (13):
  - Precision NextGen Oncology, Beverly Hills, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists-Omaha-69066, Omaha, Nebraska
  - Northwell Health, Lake Success, New York
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists Cancer Center, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Sanatorio Finochietto, CABA, Argentina
- Australia (2):
  - Prince of Wales Hospital-Randwick-66496, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Canada (2):
  - Arthur J. E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Sun Yat-Sen University Cancer Center, Guangzhou, China
- University Hospital Olomouc, Olomouc, Czechia
- Copenhagen University Hospital, Rigshospitalet, København Ø, Denmark
- France (2):
  - CTR Leon Berard, Lyon
  - CTR Eugène Marquis, Rennes
- Germany (2):
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Tübingen, Tübingen
- Clinexpert Gyongyos, Gyöngyös, Hungary
- Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (7):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Chuo-ku
- Oslo Universitetssykehus HF, Radiumhospitalet, Oslo, Norway
- Oncology Center-Maria Sklodowska-Curie Institute, Warsaw, Poland
- Spain (5):
  - Hospital Universitario Miguel Servet, Aragon
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
- Karolinska Comprehensive Cancer Center, Stockholm, Sweden
- Taipei Veterans General Hospital, Taipei, Taiwan
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - University College Hospital, London
  - The Royal Marsden Hospital, Chelsea, London

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com